CLINICAL TRIAL: NCT03672032
Title: Randomized Controlled Trial Comparing the Franseen Needle With a Fork-tip Needle for EUS-guided Fine Needle Biopsy
Brief Title: SharkCore Versus Acquire FNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Gerke (Other)
Responsible Party: Sponsor-Investigator, Henning Gerke, MD, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201808820
Record Dates: First submitted 2018-08-30; First posted 2018-09-14 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: EUS Guided Biopsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fork-tip Needle (Active Comparator)
  Interventions: Device: Fork-tip Needle
- Franseen Needle (Active Comparator)
  Interventions: Device: Franseen Needle

INTERVENTIONS:
Device: Fork-tip Needle — Fork-tip Needle will be used to obtain biopsy
  Arms: Fork-tip Needle
Device: Franseen Needle — Franseen Needle will be used to obtain biopsy
  Arms: Franseen Needle

SUMMARY:
Endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) has been established as an effective technique for sampling tissue inside and around the gastrointestinal tract, including the pancreas, liver, lymph nodes, and adrenal glands. EUS-FNA is convenient, minimally invasive, and safe procedure with an estimated sensitivity of 75%-92% and a specificity of 82%-100%.

Diagnosis of various pathologies in the GI tract including solid pancreatic masses, mediastinal or gastric lymph nodes, gastrointestinal submucosal lesions, and peri-rectal lesions require adequate tissue architecture and immunohistochemical analysis. This is difficult to obtain and is frequently insufficient with EUS-FNA cytology alone. The core tissue is required to improve the diagnostic yield and obtain histologic diagnosis along with immunostaining to establish specimen adequacy. In past 1 year two new needle EUS needle (Shark Core)and Acquire EUS needles has been introduced to improve diagnostic accuracy, tissue yield, and potentially obtain a core tissue sample. So far, no prospective studies have compared these two needles to see which one is better for overall diagnostic accuracy. Our goal is to perform a prospective analysis to compare the diagnostic yield and safety profile of these 2 new EUS needle.

DETAILED DESCRIPTION:
Subjects will come to a pre-procedure room on the day of the procedure. The investigator will again go over the risk and benefit of procedure and indication of the procedure. Once the consent form is signed, a large bore IV cannula is placed and the subject will be taken to the DHC procedure room. Once all the team members required to perform the procedure are in the room we will do a time-out to make sure current patient and procedure are performed. A time-out is done by asking the subject to tell his full name with date of birth and describe in his own words what procedure is planned for subject today. If all the things match the investigator will go ahead and start the sedation.

All EUS-FNB will be performed in the standard manner using linear echoendoscopes. All EUS-FNB procedures were performed by 1 of 2 highly experienced endosonographers (Henning Gerke or Rami EL-Abiad).

The needle to be used (SharkCore vs Acquire) will be decided based on randomization software. The needle will then be used to puncture the target lesion in standard fashion. Aspirated cellular materials will be expressed into the slide by advancing the stylet. The remainder will be expressed onto filter paper and submitted for cell block preparation. The subject's medical information including diagnosis, date of diagnosis, date of admission, blood test results, and medications received will be reviewed for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients schedule for EUS guided biopsy

Exclusion Criteria:

* Patients who had EUS-FNA for cystic fluid aspiration
* Pregnant females
* International normalized ratio >1.5 and platelet count < 50,000
* Medically unstable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Gerke, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD.

REFERENCES:
- [Derived] Ashat M, Klair JS, Rooney SL, Vishal SJ, Jensen C, Sahar N, Murali AR, El-Abiad R, Gerke H. Randomized controlled trial comparing the Franseen needle with the Fork-tip needle for EUS-guided fine-needle biopsy. Gastrointest Endosc. 2021 Jan;93(1):140-150.e2. doi: 10.1016/j.gie.2020.05.057. Epub 2020 Jun 9. PMID 32526235

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Groups:
- SharkCore Needle: SharkCore Needle: SharkCore Needle will be used to obtain biopsy
- Acquire Needle: Acquire Needle: Acquire Needle will be used to obtain biopsy
Period: Overall Study
Arm/Group | SharkCore Needle | Acquire Needle
Started | 67; 75 Lesions | 67; 75 Lesions
Completed | 67; 75 Lesions | 67; 75 Lesions
Not Completed | 0; 0 Lesions | 0; 0 Lesions

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fork-tip Needle | Franseen Needle | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.81 (12.49) | 65.90 (12.34) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 33 | 37 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 67 | 67 | 134

OUTCOME MEASURES:

1. Primary Outcome: Is the Acquire Needle Non-inferior Compared to SharkCore Needle in Histologic Yield of the Sample Obtained?
Description: A pathologist blinded to clinical information will access each Biopsy specimen for adequacy (scoring system where scores of 0 were samples with no material, 1 - sufficient material for adequate histological interpretation, low quality (total material <10x power field in length), 2 - sufficient material for adequate histological interpretation, high quality (>10x power field in length)
Time Frame: 12 months
Population: Histology Adequacy Score (0-2)
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Franseen Needle: Franseen Needle: Fransee Needle will be used to obtain biopsy
Arm/Group | Fork-tip Needle | Franseen Needle
Number analyzed (Participants) | 67 | 67
Number analyzed (Lesions) | 75 | 75
Lesions
  0, Insufficient | 3 | 4
  1, Sufficient, low quality | 10 | 14
  2, Sufficient, high quality | 62 | 57

2. Secondary Outcome: Is the Acquire Needle Non-inferior Compared to SharkCore Needle in Diagnostic Accuracy?
Description: The diagnostic accuracy was calculated considering malignant diagnoses as a true positive.
  A histological or cytological diagnosis of a neoplastic lesion will be considered correct since false-positive diagnoses have been reported to be rare if strict cytological criteria are applied.
  The criterion standard for diagnosis of benign, non-neoplastic lesion that will not undergo surgical resection will be based on a combination of clinal impression, imaging characteristics and a clinical course that was consistent with the study diagnosis.
Time Frame: 12 months
Population: Combined diagnostic accuracy
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Fork-tip Needle | Franseen Needle
Number analyzed (Participants) | 67 | 67
Number analyzed (Lesions) | 75 | 75
Lesions | 69 | 65

3. Secondary Outcome: Is the Acquire Needle Non-inferior Compared to SharkCore Needle in Number of Needle Passes Required to Obtain the Tissue Sample?
Description: We will be collecting data on how many needle passes are required to get adequate FNB sample for each procedure. In the end, we will use this data to calculate using standard statistical measures to compare the average number of passes required to get adequate sample by both SharkCore and Acquire needle.
Time Frame: 12 months
Population: Needle passes
Measure: Median (Inter-Quartile Range); unit: number of needle passes
Units Other Than Participants: Lesions
Arm/Group | Fork-tip Needle | Franseen Needle
Number analyzed (Participants) | 67 | 67
Number analyzed (Lesions) | 75 | 75
number of needle passes | 3 [2 to 4] | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Fork-tip Needle | Franseen Needle
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/67
Other Adverse Events (participants affected / at risk) | 8/67 | 9/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fork-tip Needle (N=67) | Franseen Needle (N=67)
Bleeding (Hepatobiliary disorders) | 0 (0) | 1 (1) — Small hepatic hematoma. No intervention required. Patient was discharged after 1 day.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fork-tip Needle (N=67) | Franseen Needle (N=67)
Pancreatitis (Hepatobiliary disorders) | 2 | 3
Abdominal Pain (General disorders) | 4 | 5
Nausea/Vomiting (Gastrointestinal disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT03672032/Prot_SAP_000.pdf